CLINICAL TRIAL: NCT07228247
Title: A Phase Ⅰ/Ⅱa Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of HMPL-A251 in Participants With Advanced or Metastatic HER2-Expressing Solid Tumors
Brief Title: A Phase Ⅰ/Ⅱa Study of HMPL-A251 in Participants With Advanced or Metastatic HER2-expressing Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-251-GLOB1
Record Dates: First submitted 2025-11-11; First posted 2025-11-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A(Phase I) (Experimental): Dose Escalation
  Interventions: Drug: HMPL-A251
- Part B(Phase IIa) (Experimental): Dose Expansion/Dose Optimization
  Interventions: Drug: HMPL-A251

INTERVENTIONS:
Drug: HMPL-A251 — Six dose cohorts are planned for the Dose Escalation phase; at least three participants with solid tumors will be enrolled in each dose cohort. Bayesian optimal interval design with backfill (BF-BOIN, Zhao, 2023) will be used to guide dose escalation and determine the MTD and/or RDE of HMPL-A251. All study participants will receive HMPL-A251 as IV infusion until PD, intolerable toxicity, or other protocol-specified criteria for ending study treatment, whichever occurs first.
  Arms: Part A(Phase I)
Drug: HMPL-A251 — Participants will be randomized in a 1:1 ratio to receive treatment in two RDEs levels (approximately 15 participants per dose level) for each cohort. All study participants will receive HMPL-A251 as IV infusion until PD, intolerable toxicity, or other protocol-specified criteria for ending study treatment, whichever occurs first.
  Arms: Part B(Phase IIa)

SUMMARY:
This is a first-in-human (FIH), phase Ⅰ/Ⅱa, open-label, multicenter clinical study of HMPL-A251 monotherapy in adult participants with unresectable, advanced or metastatic HER2-expressing solid tumors.

DETAILED DESCRIPTION:
* To evaluate the safety and tolerability and to determine the maximum tolerated dose (MTD) and/or recommended dose(s) for expansion (RDE) of HMPL-A251 in participants with previously treated HER2+ solid tumors
* To characterize the safety and preliminary efficacy of HMPL-A251 at RDEs to determine recommended dose(s) for phase 2 (RP2D) or phase 3 (RP3D) in participants with selected HER2-expressing solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed unresectable advanced or metastatic disease.
2. Have at least one measurable lesion per RECIST v1.1;
3. Life expectancy ≥ 12 weeks;
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1;
5. Weight ≥ 35 kg;

Exclusion Criteria:

1. An established diagnosis of type I diabetes mellitus or uncontrolled type II diabetes mellitus.
2. Use of strong inhibitors of cytochrome P450 3A4 enzyme (CYP3A4), and inhibitors of P-glycoprotein (P-gp) and breast cancer resistance protein (BCRP) within 5 elimination half-lives or 2 weeks (whichever is longer) before the first dose of study drug;
3. Toxicity from prior anti-tumor therapy has not recovered to Grade 1 or baseline prior to the first dose of study drug (except alopecia). Participants with chronic Grade 2 toxicities may be eligible after discussion between the investigator and Sponsor Medical Monitor (e.g., Grade 2 chemotherapy-induced neuropathy);
4. Baseline blood amylase or lipase exceeds the normal range and are judged by the investigators to be clinically significant;
5. Spinal cord compression, leptomeningeal disease, or clinically active central nervous system (CNS) metastases, defined as untreated or symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms;
6. Major surgery within 28 days prior to the first dose of study drug. Participants must have recovered adequately from the toxicity and/or complications from the intervention prior to the first dose of study drug(s);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Approximately 12 months
  At least three participants will be enrolled in each dose cohort. Bayesian optimal interval design with backfill (BF-BOIN) will be used to guide dose escalation and to determine the MTD of HMPL-A251
Recommended doses for expansion (RDE) | Approximately 12 months
  The RDE will be selected by evaluating all available data from the following criteria under consideration: Determination of MTD achieved during the dose escalation part; Safety data obtained across all different doses tested; Tolerability data, such as chronic toxicities, discontinuations, or withdrawals for toxicity that occur beyond the DLT period; PK data collected at the time of evaluation; Preliminary efficacy data.
Overview of Treatment-emergent Adverse Events (TEAEs) | Approximately 24 months
  All TEAEs will be graded according to NCI CTCAE v6.0 and coded using the Medical Dictionary for Regulatory Activities (MedDRA).
Objective Response Rate (ORR) | At least 6 weeks post dose of first participant up to approximately 24 months
  ORR is defined as the proportion of participants with Best objective response (BOR) of confirmed complete response (CR) or partial response (PR), as per investigator's assessment according to RECIST v1.1.
Recommended doses for phase II or III studies (RP2D or RP3D) of HMPL-A251 | Approximately 12 months
  The RP2D or RP3D will be selected by evaluating all available data from the following criteria under consideration: Determination of MTD achieved during the dose escalation part; Safety data obtained across all different doses tested; Tolerability data; PK data; efficacy data.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Approximately 2 years
  The proportion of participants with BOR of confirmed CR, confirmed PR, or stable disease (SD) lasting at least 5 weeks.
Duration of response (DoR) | Approximately 2 years
  Only applies to participants whose BOR is confirmed CR or PR and is defined as the time from the first occurrence of objective tumor response (CR or PR) to the date of first radiographic PD or death due to any cause.
Time to response (TTR) | Approximately 2 years
  Only applies to participants whose BOR is confirmed CR or PR and is defined as the time from the first dose of study dose to the first occurrence of objective tumor response (CR or PR)
Progression-free survival (PFS) | Approximately 2 years
  The time from the first dose of study drug to the date of first radiographic PD per RECIST v1.1 or death due to any cause, whichever occurs first.
Overall survival (OS) | Approximately 2 years
  Every 12 weeks (± 7 days) until death, withdrawal of consent for follow-up, lost to follow-up or end of study, whichever occurs first.
Pharmacokinetic Analysis(Cmax) | Each cycle(21-day cycle), From C9, every 4 cycles, Approximately 12 months
  Maximum Observed Serum Concentration
Pharmacokinetic Analysis(Tmax) | Each cycle(21-day cycle), From C9, every 4 cycles, Approximately 12 months
  Time to Peak Plasma Concentration
Pharmacokinetic Analysis((AUC) | Each cycle(21-day cycle), From C9, every 4 cycles, Approximately 12 months
  Area Under the Concentration Versus Time Curve
To evaluate the immunogenicity of HMPL-A251 | Each cycle(21-day cycle), From C9, every 4 cycles, Approximately 12 months
  Incidence of anti-drug antibody and neutralizing antibody against HMPL-A251

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - SCRI HealthONE, Denver, Colorado
  - BRCR Global, Plantation, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
- China (6):
  - Peking University First Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - Fujian Cancer Hospital, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Henan Cancer Hospital, Zhengzhou